CLINICAL TRIAL: NCT01915550
Title: The Role of Adding Metformin in Insulin-Resistant Diabetic Pregnant Women - a Randomized Controlled Trial
Brief Title: Metformin as Adjuvant to Insulin Therapy in Insulin-resistant Diabetes Mellitus With Pregnancy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohammed Faris, Assistant Lecturer of Obstetrics and Gynecology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 361979
Record Dates: First submitted 2013-08-02; First posted 2013-08-05 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2013-08

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes mellitus; Pregnancy; Insulin; Metformin
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance | interventions — Metformin

ARMS (2):
- metformin (Active Comparator): metformin was added without raising the insulin dose
  Interventions: Drug: Metformin
- Raising Insulin (Active Comparator): insulin dose is raised
  Interventions: Drug: Humulin Insulin Mixtard

INTERVENTIONS:
Drug: Metformin
  Other Names: Cidophage
  Arms: metformin
Drug: Humulin Insulin Mixtard
  Arms: Raising Insulin

SUMMARY:
Adding metformin to insulin therapy in pregnant women with diabetes mellitus who show insulin resistance may be equivalently effective to further raising the insulin dose

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with insulin-resistant diabetes mellitus

Exclusion Criteria:

* type-1 diabetes mellitus
* secondary diabetes mellitus

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2012-04; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Proper Glycemic Control | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Cairo Governorate, Egypt